CLINICAL TRIAL: NCT05359601
Title: Effect of Infusion Set Replacement Intervals on Central Line-associated Bloodstream Infection in Adult Intensive Care Unit: a Multicenter Randomised Clinical Trial
Brief Title: Infusion Set Replacement Intervals for Critically Ill Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BHu
Record Dates: First submitted 2022-03-28; First posted 2022-05-04 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Critical Illness
Keywords: Infusion set; CLABSI; Intensive care unit; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24-hour (Experimental): Every 24-hour infusion set replacement
  Interventions: Procedure: Infusion set replacement intervals
- 96-hour (Placebo Comparator): Every 96-hour infusion set replacement
  Interventions: Procedure: Infusion set replacement intervals

INTERVENTIONS:
Procedure: Infusion set replacement intervals — 24-hour or 96-hour infusion set replacement intervals

SUMMARY:
This study aimed to evaluate the efficacy of 24-hour versus 96-hour infusion set replacement to prevent central line-associated bloodstream infection (CLABSI) in critically ill adults with central venous access devices.

DETAILED DESCRIPTION:
Up to 70% of patients in acute care hospitals need a central venous access, and the latter is also widely used in other clinical settings. However, the central venous access usually remains associated with increased infection risks, which can be severe and even lethal.

Most contemporary guidelines recommend infusion set replacement every 4 days with the CDC in US recommending replacement "no more frequently than 96 hours, but at least every 7 days". However, the National Health Commission of the People's Republic of China recommend infusion set replacement every 24 hours in 2021. The previous evidence from neonate were in favor of the administration set changes of every 24 hours, compared with the longer time interval. However, it is unclear whether this conclusion applied to adult critically ill patients in ICU.

The purpose of the current study is therefore to compare the effectiveness of 24-hour versus 96-hours infusion set replacement to prevent central line-associated bloodstream infection (CLABSI) in critically ill adults with central venous access devices.

This study is a multicenter, single-blind randomized clinical trial designed to investigate the efficacy of the 24-hour versus 96-hours infusion set replacement to prevent central line-associated bloodstream infection (CLABSI) in critically ill adults with central venous access devices. The trial will enroll up to 1240 participant. The primary endpoint for this trial is the CLABSI rate. Mortality rate is a key secondary endpoint for the trial.

Specific Aims

1. To demonstrate the efficacy of 24-hour infusion set replacement to reduce the rate of CLABSI, compared with 96-hours infusion set replacement.
2. To demonstrate the efficacy of 24-hour infusion set replacement to reduce the rate of CRBSI, all-cause bloodstream infection, and mortality, compared with 96-hours infusion set replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Able to provide informed consent
3. Expected length of stay (LOS) > 96 hours in intensive care unit (ICU)
4. Need for treatment with central venous access device
5. The central venous access device is expected to remain in place for at least 96 hours, with infusion set attached

Exclusion Criteria:

1. Those who with a bloodstream infection within the previous 48 hours after ICU admission
2. Those who have their vascular access device actually removed within 96 hours after ICU admission
3. Those who have participated in other clinical studies within the 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Central-line associated bloodstream infections (CLABSI) rates | Day 28
  i) the catheter was in place for at least 48 hours prior to onset of sepsis, and/or ii) there was microbiologic growth (bacteria and/or fungi) of at least 15 colony forming units (CFU) on the CVC tip identical to a positive blood culture sample, and/or iii) the difference in time to positivity between a central and a peripheral drawn blood culture was more than 2 hours

SECONDARY OUTCOMES:
Catheter-related bloodstream infection (CRBSI) rates | Day 28
  A bacteraemia or fungaemia (with clinical manifestations of infection and no other identifiable source) and at least one positive blood culture from a peripheral vein, plus matching organism(s) found on the catheter tip (>15 CFUs on semiquantitative culture); or, two blood cultures (one from catheter, one from peripheral vein) with matching organism(s) that met the criteria for differential time to positivity (growth of catheter-drawn blood at least 2 h before growth from a peripheral vein blood culture)
All-cause bloodstream infection rates | Day 28
  All-cause bloodstream infection
Colonisation of vascular access device | Day 4
  Semiquantitative method ('Maki roll'), cutoff ≥15 cfu/catheter
Colonisation of infusion set | Day 4
  Quantitative (broth dilution) method, cutoff ≥1000 cfu/ml
ICU all-cause mortality | Day 28
  Number of patients who were confirmed to be dead in ICU from enrollment onto the study
In-hospital all-cause mortality | Day 28
  Number of patients who were confirmed to be dead in hospital from enrollment onto the study
28-day all-cause mortality | Day 28
  Number of patients who were confirmed to be dead within 28-day from enrollment onto the study
ICU length of stay | Day 28
  Length of intensive care unit stay
Hospital length of stay | Day 28
  Length of hospital stay
The cumulative time of catheter in situ | Day 28
  The cumulative time of catheter in situ
The number of infusion sets used per patient | Day 28
  The cumulative number of individual infusion sets used per patient
The costs of consumables for doing all infusion set replacement procedures per patient | Day 28
  The cumulative costs of consumables for doing all infusion set replacement procedures per patient
The cumulative staff time for doing all infusion set replacement procedures per patient | Day 28
  The cumulative staff time for doing all infusion set replacement procedures per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu D, Hu C, Xiong J, Huang H, Wang S, Ding X, Zhou J, Deng J, Guo C, Li M, You T, Cheng W, Li B, Tang X, Li X, Li H, Li J, Ma J, Xiao M, Fu X, Li H, Peng Z, Hu B, Hu F; INSPIRATION Study group. Effect of Infusion Set Replacement Intervals on Central Line-Associated Bloodstream Infection in the Intensive Care Unit: Study Protocol of the INSPIRATION Study. Infect Dis Ther. 2024 Apr;13(4):941-951. doi: 10.1007/s40121-024-00953-y. Epub 2024 Mar 14. PMID 38483776